CLINICAL TRIAL: NCT02523352
Title: Evaluation of Effects of Positive End-expiratory Pressure (PEEP) on Lung and Heart Functions in Spontaneous Breathing Obese Subjects.
Brief Title: Effects of PEEP on Heart and Lungs in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, RRT, PhD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EIT-TTE-MRI-Obese
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Pulmonary Atelectasis; Obesity Hypoventilation Syndrome; Magnetic Resonance Imaging; Respiratory Mechanics; Electrical Impedance Tomography; Trans-Thoracic Echocardiography
MeSH Terms: conditions — Obesity; Pulmonary Atelectasis; Obesity Hypoventilation Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: 35 patients will be enrolled in this study. The study is divided in two phases: the first phase will evaluate the PEEP in 12 consecutive obese subjects and 6 healthy volunteers using Trans-thoracic echocardiography (TTE) and Electrical Impedance Tomography (EIT). The second phase will evaluate the PEEP in the other 12 consecutive obese subjects and 5 healthy volunteers using Magnetic Resonance Imaging (MRI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Volunteers with a BMI > 35 Kg/m2 and central fat distribution, without any past medical history
  Interventions: Procedure: Non-Invasive Ventilation; Procedure: Esophageal catheter positioning

INTERVENTIONS:
Procedure: Non-Invasive Ventilation — Progressive increase in airway pressure to open lungs atelectatic regions.
Procedure: Esophageal catheter positioning — The esophageal tube (8 French diameter catheter) will be positioned in the larger nostril previous topical anesthesia

SUMMARY:
Aim of this study is to better understand pathophysiology of the alteration of respiratory mechanics and cardiovascular function in obese volunteer subjects. The investigators plan to test this hypothesis with a physiological, interventional study conducted on volunteers by using Electrical Impedance Tomography in a group of patients and magnetic resonance imaging (MRI) in another group.

DETAILED DESCRIPTION:
Obese subjects are prone to develop respiratory insufficiency when requiring mechanical ventilation. Atelectasis is the primary responsible for respiratory insufficiency and impossibility to wean obese patients from respiratory support. The investigators do believe that the respiratory system derangements observed in the previous study during the critical illness are already present, although in lower severity, in the obese patients in their basal condition.

This study will help to understand the standard cardiac and respiratory function of an obese non critically ill subject to better target the therapies during the management of the critical illness to reestablish the homeostasis of the system:

The investigator's hypotheses are:

* To demonstrate if morbidly obese patients show atelectasis at spontaneous breathing in the supine position and whether the increase in lung volume following PEEP titration is due to alveolar recruitment rather than overdistention.
* To measure regional variations in ventilation/perfusion coupling at different ventilator settings
* To investigate the role of diaphragm position in the development/treatment of respiratory insufficiency due to increased pleural pressure
* To test if reopening of lung atelectasis through the application o a recruitment maneuver and titrated PEEP level would lead to an improvement in right heart function.
* To assess pulmonary circulation at different levels of PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Have a photo identification document
* BMI ≥ 35 kg/m2
* Waist circumference > 88 cm (for women)
* Waist circumference > 102 cm (for men)

Exclusion Criteria:

* Psychiatric disturbances such as anxiety, depression, schizophrenia requiring pharmacological treatment or hospitalization in the last year
* Subjects with any known condition, including claustrophobia or pain, which limits their ability to lie in the MR scanner for the duration of the research study
* Known presence of esophageal varices
* Recent esophageal trauma or surgery
* Known Coagulopathy
* History of pneumothorax
* Pregnancy
* Diabetes
* Presence of prosthesis incompatible with MR
* Thoracic diameter grater than 70 cm
* Resting heart rate (HR) < 50 or > 120 bpm and/or systolic blood pressure < 90 or > 160 mmHg and/or peripheral oxygen saturation (SpO2) < 88%
* Currently enrolled in another research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
End Expiratory Lung Volume | Change from baseline [0 PEEP] to titrated PEEP level (30 minutes after baseline)
  Difference in end expiratory lung volume measured in mL

SECONDARY OUTCOMES:
Work of breathing | Change from baseline [0 PEEP] to titrated PEEP level (30 minutes after baseline)
  Difference in work of breathing will be measured as Joule/min
Right heart volumes | Change from baseline [0 PEEP] at titrated PEEP level (30 minutes after baseline)
  Difference in right heart and diastolic and end systolic volumes will be measured
Heart ejection fraction | Changes from baseline [0 PEEP] at titrated PEEP level (30 minutes after baseline)
  Difference in heart ejection fraction will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, RRT, PhD, Principal Investigator — Massachussets General Hospital; Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Behazin N, Jones SB, Cohen RI, Loring SH. Respiratory restriction and elevated pleural and esophageal pressures in morbid obesity. J Appl Physiol (1985). 2010 Jan;108(1):212-8. doi: 10.1152/japplphysiol.91356.2008. Epub 2009 Nov 12. PMID 19910329
- [Background] Chahal H, McClelland RL, Tandri H, Jain A, Turkbey EB, Hundley WG, Barr RG, Kizer J, Lima JAC, Bluemke DA, Kawut SM. Obesity and right ventricular structure and function: the MESA-Right Ventricle Study. Chest. 2012 Feb;141(2):388-395. doi: 10.1378/chest.11-0172. Epub 2011 Aug 25. PMID 21868467
- [Background] Steier J, Lunt A, Hart N, Polkey MI, Moxham J. Observational study of the effect of obesity on lung volumes. Thorax. 2014 Aug;69(8):752-9. doi: 10.1136/thoraxjnl-2014-205148. Epub 2014 Apr 15. PMID 24736287
- [Background] Tedjasaputra V, Sa RC, Arai TJ, Holverda S, Theilmann RJ, Chen WT, Wagner PD, Davis CK, Kim Prisk G, Hopkins SR. The heterogeneity of regional specific ventilation is unchanged following heavy exercise in athletes. J Appl Physiol (1985). 2013 Jul 1;115(1):126-35. doi: 10.1152/japplphysiol.00778.2012. Epub 2013 May 2. PMID 23640585
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Derived] Florio G, De Santis Santiago RR, Fumagalli J, Imber DA, Marrazzo F, Sonny A, Bagchi A, Fitch AK, Anekwe CV, Amato MBP, Arora P, Kacmarek RM, Berra L. Pleural Pressure Targeted Positive Airway Pressure Improves Cardiopulmonary Function in Spontaneously Breathing Patients With Obesity. Chest. 2021 Jun;159(6):2373-2383. doi: 10.1016/j.chest.2021.01.055. Epub 2021 May 8. PMID 34099131